CLINICAL TRIAL: NCT06499480
Title: Italian Registry of Patients With Allergic Disease and Treated With Allergen ImmunoTherapy
Brief Title: Italian Registry of Allergen ImmunoTherapy
Acronym: RIAIT
Status: Recruiting | Type: Observational
Sponsor: Società Italiana di Allergologia, Asma e Immunologia Clinica (Other)
Collaborators: Società Italiana di Allergologia e Immunologia Pediatrica (SIAIP) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2732
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Allergic Respiratory Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
RIAIT (Italian Registry of Allergy Immunotherapy) is a multicenter observational study that aims to prospectively collect the most extensive data available on Italian patients using AIT for respiratory allergies (rhinoconjunctivitis and/or asthma) in a real-life context, through a network of allergy centers with specific interest and expertise in the management of allergic respiratory patients.

DETAILED DESCRIPTION:
Objectives include:

* Evaluate short and long-term real-life effectiveness and safety of AIT overall, in specific patient groups' phenotypes and with specific AIT products.
* Evaluate the pertinence and differences in suggesting AIT to a patient comparing physician's evaluation in various settings with established international guidelines, describing the factors associated with treatment choices and changing over time, and promoting interoperability, data sharing, and cross-comparison among centers.
* Describe long-term respiratory allergic disease evolution in patients treated with AIT.
* Describe the natural history of the patient population with respiratory allergies and identify patient groups describing their illness burden, management patterns, and clinical progression.
* Promote the creation of accurate, standardized, and efficient processes for diagnosing and treating respiratory allergic diseases, especially with AIT.
* Assess biomarker data to predict diagnosis, treatment response and long-term disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 year
* Confirmed diagnosis of allergic rhinoconjunctivitis and/or allergic asthma according to EAACI 2019 guidelines.
* Having been followed by the recruiting center for at least one month: this is considered necessary to establish that the patients are truly affected by allergic respiratory disease and are eligible for allergen-specific immunotherapy; in this period, screening tests are carried out to exclude and/or confirm concomitant diseases (comorbidities). In fact, according to the aforementioned EAACI guidelines, a patient can be defined as truly eligible for allergen-specific immunotherapy only after a preliminary phase in which the patient is treated with symptomatic therapy; this observation period allows a correct evaluation of the real adherence and response to therapy, as well as the identification and appropriate treatment of any comorbidity and the possible elimination of aggravating factors.
* Having received the prescription of any of the available AIT products in Italy, irrespectively of the selected allergens and the administration route and schedule.

Exclusion Criteria:

There will no be exclusion criteria, in order to allow a real-life vision of the characteristics of these patients eligible for or treated with allergen-specific immunotherapy.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RIAIT is a prospective multicenter observational registry of patients suffering from conjunctivitis, rhinitis, and/or allergic asthma eligible for and treated with AIT according to EAACI (European Academy of Allergy and Clinical Immunology) Guidelines.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Life Quality as measured by Standardised Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ(S)) (≥12years) | Every year to ten year
Life Quality as measured by Paediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) For Children 6 - 12 years | Every year to ten year

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Marco Heffler, MD, PhD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (2):
- Italy (2):
  - Personalized Medicine, Asthma and Allergy - IRCCS Humanitas Research Hospital, Rozzano, Italy, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Istituto di Ricovero e Cura a Carattere Scientifico, Florence